CLINICAL TRIAL: NCT06126055
Title: EndoBand: Endoscopic Band Ligation for Treating Reflux Disease (GERD)
Brief Title: Endoscopic Band Ligation for Treating Reflux Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: El Katib Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abeid, Consultant Gastroenterologist, El Katib Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIELUKA
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: GERD
Keywords: GERD; GastroEsophageal Reflux; Band Ligation; EndoBand
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Off PPI (Experimental): No symptoms of reflux
  Interventions: Device: Band Ligation

INTERVENTIONS:
Device: Band Ligation — Placing bands in distal esophagus

SUMMARY:
GERD is a chronic disease the require different treatment modalities; non have proven long term efficacy with concerns about their safety. The use of band ligation in endoscopy appears safe, repeatable with short learning curve. Placing multiple bands at the Z-line can create a fibrous ring in the distal esophagus acting as a barrier against reflux of gastric content.

DETAILED DESCRIPTION:
The aim of the study is the complete resolution of reflux symptoms without the use of any drug.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic GERD

Exclusion Criteria:

* Any previous surgery for GERD

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic Band Ligation for GERD | 1 month
  Resolution of reflux symptoms and stopping proton pump inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abeid, MD, Principal Investigator — Endoscopy Unit Faculty of Medicine Cairo University
Locations (1):
- Endoscopy Unit Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Free
URL: http://www.MohamedAbeid.com